CLINICAL TRIAL: NCT01240655
Title: A Phase Ib Study of LCL161 in Combination With Weekly Paclitaxel in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of LCL161 in Combination With Weekly Paclitaxel in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCL161A2104; 2009-015594-12 (EudraCT Number)
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-09

CONDITIONS: Solid Tumors
Keywords: LCL161; solid tumors; paclitaxel
MeSH Terms: interventions — LCL161; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCL161 + Paclitaxel (Experimental)
  Interventions: Drug: LCL161; Drug: Paclitaxel

INTERVENTIONS:
Drug: LCL161
Drug: Paclitaxel

SUMMARY:
This is a dose escalation study that will assess the safety and efficacy of LCL161 in combination with weekly paclitaxel in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Patients with breast cancer must have a histologically or cytologically confirmed diagnosis of disease that has metastasized or is resistant to therapy.

Patients with ovarian cancer must have histological evidence of recurrent epithelial ovarian, fallopian tube or peritoneal cancer.

Patients must have recovered or stabilized from all toxicities related to their previous treatment except for alopecia Male or female patients 18 years or older ECOG performance status 0-1 Life expectancy greater than 12 weeks Measurable disease as determined by RECIST v1.0 Patients must give written informed consent and comply with the protocol

Exclusion Criteria:

For patients with breast cancer:

Concurrent Her2-directed or anti-estrogen therapy

For patients with ovarian cancer:

Primary refractory disease, defined as progression during initial treatment with a platinum- and taxane-containing regimen.

Prior treatment with weekly paclitaxel. More than two chemotherapy regimens given in the relapse setting. Evidence of a documented bowel obstruction within six months of study entry Patients with unresolved peripheral neuropathy, nausea, vomiting, or diarrhea ≥ CTCAE Grade 2 Any concurrent severe and/or uncontrolled medical conditions that could increase the patient's risk for toxicity while in the study or that could confound discrimination between disease- and study treatment-related toxicities.

Patients with impairment of GI function or GI disease that may significantly alter the absorption of LCL161 Patients who have undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of procedure.

Pregnant or breast feeding (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive β-HCG laboratory test (> 5 mIU/mL).

Known diagnosis of human immunodeficiency virus (HIV) infection or chronic active hepatitis B or C (HIV and hepatitis testing are not mandatory).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD)/RP2D of LCL161 when administered in combination with once weekly paclitaxel | 24 months

SECONDARY OUTCOMES:
Safety and tolerability of the combination, including acute and chronic toxicities | 24 months
Pharmacokinetics of both LCL161 and paclitaxel when administered in combination (AUC0-∞, Cmax, tmax and other parameters as appropriate) | 24 months
Preliminary anti-tumor activity associated with this combination treatment | 24 months
Target inhibition, cell death, and cytokines in surrogate and tumor tissues | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (3):
  - Dana Farber Cancer Institute SC, Boston, Massachusetts
  - University of North Carolina Lineberger Comp Cancer Ctr, Chapel Hill, North Carolina
  - Sarah Cannon Research Institute DeptofSarahCannonRes.Inst. (2), Nashville, Tennessee
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- Novartis Investigative Site, Modena, MO, Italy
- Novartis Investigative Site, Barcelona, Catalonia, Spain

REFERENCES:
- See also: Results for CLCL161A2104can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14450